CLINICAL TRIAL: NCT05547295
Title: Evaluation of the Impact of a Digital Tool MEDIASCREEN of Preventive Information for Patients on the Knowledge of the Risk of Pressure Sores Acquired During a Hospitalization, a Randomized Controlled Pilot Interventional Study in Single Blind
Brief Title: Evaluation of the Impact of a Digital Tool MEDIASCREEN of Preventive Information for Patients on the Knowledge of the Risk of Pressure Sores Acquired During a Hospitalization
Acronym: EDUCESCARRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-A00520-43
Record Dates: First submitted 2022-07-07; First posted 2022-09-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pressure Sore
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper Information (Other): Patient will have classic paper information for prevention of pressure sores
  Interventions: Other: Paper prevention
- Numeric information from MEDIASCREEN (Experimental): Patient will have information for prevention of pressure sores throught the digital tool MEDIASCREEN
  Interventions: Other: Numeric prevention

INTERVENTIONS:
Other: Numeric prevention — Numeric information for prevention of pressure sores thgrough digital tool MEDIASCREEN
  Arms: Numeric information from MEDIASCREEN
Other: Paper prevention — Information for prevention of pressure sores in classic way with paper
  Arms: Paper Information

SUMMARY:
The study focuses on the impact of a digital MEDIASCREEN tool on the knowledge, technical know-how and behavioural skills in terms of pressure sores of patients. In addition, the cognitive impact of this type of tool will also be studied in our study population (self-esteem and feeling of personal effectiveness). The objective is to compare the impact of a digital MEDIASCREEN information tool with information tool compared to the usual paper-based prevention materials on knowledge of the risk of hospital-acquired pressure sores.

ELIGIBILITY:
Inclusion Criteria:

* Patient in complete hospitalization in Physical Medicine and Rehabilitation
* Patient affiliated to a social security system
* Patient presenting a low to high risk of pressure ulcer inferior or equal to or equal to 16 on the Norton scale
* Patient having signed his consent

Exclusion Criteria:

* Difficulty understanding and is unable to give free and informed consent
* Pregnant women
* Person deprived of liberty by a judicial or administrative administrative decision
* Major under legal protection by a judicial or administrative decision.
* Person in an emergency situation unable to give their informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Evaluate the change on the knowledge of the risk of hospital-acquired pressure sores with a digital MEDIASCREEN information tool in comparison to the usual paper-based prevention materials | Change from baseline knowledge at 1 month
  The comparison will be done with Skin-Management Needs Assessment Checklist score (SMNac). Minimum value =0, Maximum value = 100; higher score better outcome.

SECONDARY OUTCOMES:
Evaluate patient satisfaction with the information delivered by the MEDIASCREEN digital tool | At 1 month
  Measured by Visual Analogic scale from 0 to 100. Zero is represented : "Not at all satisfied" and 100 : "Completely satisfied".
  Higher scores better outcome.
Assess the cognitive impact of the prevention information delivered by MEDIASCREEN tool, on self-esteem. | At the beginning and at 1 month
  Measured of self-esteem with Rosenberg scale. Score range : 10-40. High scores indicate high self esteem.
Assess the cognitive impact of the prevention information delivered by MEDIASCREEN tool, on sense of self-efficacy. | At the beginning and at 1 month
  Measured of self-efficacy with scale to evaluate the feeling of personal effectiveness (MSES) Score range: 16-80. High scores indicate high feeling of personal effectiveness.
Evaluate the psychological impact of information delivered from the tools | At 1 month
  Measured by Visual Analogic scale from 0 to 100. Zero is represented : "No knowledge" and 100 : "Perfectly mastered subject".
  Higher scores better outcome.
Evaluate the occurrence of pressure sores during hospitalization | At the beginning and at 1 month
  Count of the apparition number of pressure sores.
Evaluate the acquisition of knowledge by patients | At 1 month
  Evaluate with questionnaire of knowledge, compose by 5 questions on three points each. The overall questionnaire will be on 15 points.
  Higher scores better outcome.
Evaluate the user experience when using the digital tool MEDIASCREEN. | At 1 month
  Measured by Questionnaire Attrakdiff for the user experience. The AttrakDiff questionnaire contains 28 question with 7 Likert-type scale from -3 to 3.
Evaluate the observance when using the digital tool MEDIASCREEN. | At 1 month
  Measured by the connexion data : number of connexion, duration of connexion, percentage of completion.
Evaluate the acceptability of the digital information tool MEDIASCREEN digital information tool or the paper information brochure. | At the beggining and at 1 month
  The acceptability will be assessed using a 13-item questionnaire based on the Unified Theory of Acceptance and Use of Technology (UTAUT) model. Each question is based on a Likert-type 5 point scale ranging from : 1=In total disagreement, 2= Somewhat disagree, 3= Neither agree nor disagree, 4= Somewhat agree, 5=In total agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Duruflé, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pôle Saint-Hélier, Rennes, Brittany Region, France